CLINICAL TRIAL: NCT02504879
Title: Study of the Natural History, Pathogenesis and Outcome of Melorheostosis - a Rare Osteosclerotic Disease
Brief Title: Natural History, Pathogenesis and Outcome of Melorheostosis A Rare Osteosclerotic Disease
Status: Recruiting | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150165; 15-AR-0165
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01-12

CONDITIONS: Rheumatic Disease
Keywords: Osteosclerosis; Hyperostosis; Natural History
MeSH Terms: conditions — Rheumatic Diseases; Osteosclerosis; Hyperostosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Melorheostosis patients: Patients aged > 18 years with possible and confirmed melorheostosis.
- Relatives of patients with melorheostosis: Relatives of patients with melorheostosis may be included for genetic testing only.

SUMMARY:
Background:

- The rare disease melorheostosis causes bones to thicken. This may lead to pain, and can affect bones, joints, and muscles. Researchers want to learn more about the disease and how it progresses.

Objective:

-To see what happens to people with melorheostosis over time and understand the causes of the disease.

Eligibility:

* People 18 and over with melorheostosis.
* Their unaffected relatives.

Design:

* All participants will have a medical history and physical exam.
* Participants who are relatives will give samples of blood or cheek cells.
* Other participants will be in the study for about 1 week.
* They will have blood and urine collected.
* Strength, walking, and range of motion will be measured.
* Participants may also have
* X-rays and scans.
* A pain and neurological evaluation.
* Their skin evaluated by a dermatologist.
* A small sample of bone taken.
* Nerve conduction studies. Small electrodes with to wires will be put on the skin. A metal probe will give a small electrical shock.
* Electromyography. A thin needle will be placed into the muscles.
* An ultrasound, which uses sound waves to examine the muscles and nerves. An ultrasound probe will be placed over the skin.
* A bone scan. They will get a small amount of radioactive fluid through a needle in an arm vein. This fluid travels to the bones. The bones will be photographed in a machine.
* Bone Densitometry, a low-level x-ray.
* Photographs taken.
* A small circle of skin removed with a surgical instrument.
* Questionnaires about their quality of life.
* Participants will be asked to return about every 2 years. At these visits, participants may have blood and urine tests and x-rays.

DETAILED DESCRIPTION:
Melorheostosis is a rare osteosclerotic disease resulting in exuberant excessive bone growth with a characteristic radiographic appearance often described as dripping candle wax. As a result of these bony formations, patients report mild-moderate pain that interferes with their routine activities. It is usually diagnosed on radiographs but bone biopsy may be performed to exclude other osteosclerotic diseases and/or osteosarcoma. Deformities, limb-length discrepancy, muscle atrophy, neurological deficit have been reported as complications. A subset of patients have somatic mutations in MAP2K1.

The cause of this disease is not known in all patients, the natural history poorly described and there is no clearly-defined systemic therapy. We propose a prospective observational study to investigate the natural history and pathogenesis of the disease. Subjects will undergo standardized initial evaluation and medically indicated testing. Skin biopsies may be performed to test for known mutations related to melorheotosis, and if negative affected bone and/or skin may be sent for genetic testing for acquired somatic mutations in genes that control bone homeostasis. Enrolled subjects will be followed every two to three years for assessment of disease progression and receive testing and treatment. The study of this rare bone disease offers the potential to generate new insights, provide answers as well as generate new questions into the biology of the skeletal and mineral metabolism.

ELIGIBILITY:
* INCLUSION CRITERIA:

All eligible patients are invited to participate in this protocol. Patients are adults aged > 18 years with possible melorheostosis (suspected or confirmed). Since both men and women are affected with the disease, both sexes will be studied. All ethnic and racial groups are at risk and will be included.

Relatives of patients with melorheostosis may be included for genetic testing only.

EXCLUSION CRITERIA:

* Pregnant or lactating women. A pregnancy test is performed in women of childbearing potential (up to age 55) unless they have a history of hysterectomy or tubal ligation.
* Children (age less than 18 years) are excluded.
* Subjects with severe active infection or other co-morbidities that in the opinion of the investigator would warrant exclusion.
* Subjects unable to provide informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged > 18 years with possible melorheostosis. Relatives of patients with melorheostosis may be included for genetic testing only
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2015-08-16 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Disease progression | end of the study
  explore etiology and natural history of melorheostosis. Besides MAP2K1, what other genetic changes play a role in the etiology of melorheostosis. Does the disease progress to involve new bones or extend into soft tissues over time or is it static

SECONDARY OUTCOMES:
Identify medication that affect melorheostosis | end of the study
  What medications are most effective to help with pain management in melorheostosis
Identify biomarkers | end of the study
  Can biomarkers of disease activity be ascertained.

CONTACTS AND LOCATIONS:
Overall Officials: Sarthak Gupta, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Protocol is silent about IPD sharing

REFERENCES:
- [Background] Faruqi T, Dhawan N, Bahl J, Gupta V, Vohra S, Tu K, Abdelmagid SM. Molecular, phenotypic aspects and therapeutic horizons of rare genetic bone disorders. Biomed Res Int. 2014;2014:670842. doi: 10.1155/2014/670842. Epub 2014 Oct 22. PMID 25530967
- [Background] Ihde LL, Forrester DM, Gottsegen CJ, Masih S, Patel DB, Vachon LA, White EA, Matcuk GR Jr. Sclerosing bone dysplasias: review and differentiation from other causes of osteosclerosis. Radiographics. 2011 Nov-Dec;31(7):1865-82. doi: 10.1148/rg.317115093. PMID 22084176
- [Background] Jain VK, Arya RK, Bharadwaj M, Kumar S. Melorheostosis: clinicopathological features, diagnosis, and management. Orthopedics. 2009 Jul;32(7):512. doi: 10.3928/01477447-20090527-20. PMID 19634844
- [Derived] Farrell K, Comis LE, Casimir MM, Hodsdon B, Jimenez-Silva R, Dunigan T, Bhattacharyya T, Jha S. Occupational engagement, fatigue, and upper and lower extremity abilities in persons with melorheostosis. PM R. 2023 May;15(5):587-595. doi: 10.1002/pmrj.12817. Epub 2022 May 30. PMID 35403375
- [Derived] Jha S, Fratzl-Zelman N, Roschger P, Papadakis GZ, Cowen EW, Kang H, Lehky TJ, Alter K, Deng Z, Ivovic A, Flynn L, Reynolds JC, Dasgupta A, Miettinen M, Lange E, Katz J, Klaushofer K, Marini JC, Siegel RM, Bhattacharyya T. Distinct Clinical and Pathological Features of Melorheostosis Associated With Somatic MAP2K1 Mutations. J Bone Miner Res. 2019 Jan;34(1):145-156. doi: 10.1002/jbmr.3577. Epub 2018 Sep 14. PMID 30138550
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-AR-0165.html